CLINICAL TRIAL: NCT06521021
Title: CHOICE to AVOID or RESIST: Evaluating Participants' Choice of Self-regulatory Strategy on Weight Management Outcomes: A Pilot Study.
Brief Title: CHOICE to AVOID or RESIST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Riverside (Other); Northeastern University (Other); WW International Inc (Industry); The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Sarah Salvy, Professor of Medicine, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003315
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WW + Home modification and grocery delivery (AVOID) (Other): WW + modification of home food environment + online grocery shopping and delivery
  Arm assignment is selected by participant.
  Interventions: Behavioral: AVOID
- WW + Inhibitory control training (RESIST) (Other): WW + daily gamified inhibitory control training
  Arm assignment is selected by participant.
  Interventions: Behavioral: RESIST

INTERVENTIONS:
Behavioral: AVOID — Behavioral: Home food environment and grocery delivery (AVOID) Participants will receive coaching (Zoom and/or email/text) to modify their home food environment and alter cues to promote healthy food choices
  Behavioral: WW Participants assigned to all arms will receive of coaching (Zoom and/or email/text) and commercially-available weight management program focusing on diet, physical activity and mindset skills.
  Arms: WW + Home modification and grocery delivery (AVOID)
Behavioral: RESIST — Behavioral: Inhibitory control training (RESIST) Participants assigned to RESIST will receive coaching (Zoom and/or email/text) and gamified inhibitory control training.
  Behavioral: WW Participants assigned to all arms will receive coaching (Zoom and/or email/text) and commercially-available weight management program focusing on diet, physical activity and mindset skills.
  Arms: WW + Inhibitory control training (RESIST)

SUMMARY:
This trials will formally test whether participants' active choice of self-regulatory strategies (AVOID or RESIST) leads to greater adherence to weight management strategies by comparing the CHOICE arms to the randomized arms of the parent intervention, AVOID/RESIST (IRB STUDY00001652: AVOID-RESIST).

DETAILED DESCRIPTION:
Since we initiated recruitment for the AVOID/RESIST trial (IRB STUDY00001652: AVOID-RESIST), we have noted that some participants have a strong initial inclination for one of the self-regulatory strategies. Some individuals have clearly expressed which strategy they believed would work for them, while others have voiced dislike or skepticism for an assigned intervention component. While attrition in the last 18 months (12.5%) is comparable to trials of similar size and scope, over 56% (n=18) of withdrawals were explicitly (n=3) or tangentially (n=15) related to intervention assignment.

This pilot study (CHOICE) seeks to leverage our ongoing R01 to test whether participants' active choice of behavior change pathways and strategies leads to better adherence, retention, and engagement. Consistent with ongoing procedures, women, and men with overweight or obesity (BMI between 25-45 kg/m2) will be enrolled in the WW digital program for 12 months. R01 participants will continue to be randomized to one of the 4 study arms: (1) WW alone, (2) WW + AVOID, (3) WW + RESIST, (4) WW + AVOID + RESIST. CHOICE participants will be asked to choose which self-regulatory strategy (AVOID or RESIST) they want to receive to promote behavior change consistent with WW recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* BMI between 25-45 kg/m2
* Read, write, and speak English with acceptable visual acuity

Exclusion Criteria:

* Currently enrolled in weight loss interventions or undergoing bariatric surgery
* Pregnant women
* Individuals for whom weight loss may be contraindicated (e.g., unstable coronary artery disease, end-stage disease, active cancer treatment, uncontrolled insulin-dependent diabetes, portal hypertension, drug/alcohol abuse)
* Individuals who have pacemakers or other electronic medical device implantations
* Individuals with severe cognitive delays or visual/hearing impairment
* Individuals who are unable or unwilling to complete the study assessments / measurements
* Individuals currently subscribed to a meal delivery service who are unwilling to pause their subscription for the duration of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Follow-up Completion | Baseline, 6 Month, 12 Month
  We will continuously track the rate of 6- and 12-month follow-up completion as followed: actual follow-ups completed / expected follow-ups to be completed.

SECONDARY OUTCOMES:
Height | Baseline
  Participant baseline height is self-reported in inches.
Demographics | Baseline
  Demographic questionnaire will be used to capture date of birth, sex and gender identity, race, ethnicity, socioeconomic status (education, household income, marital status, employment status) and household composition (e.g., multigenerational, children).
Drivers of preference, retention, and adherence | Baseline, 6 Month, 12 Month
  Our quantitative analytic approach will make it possible to compare CHOICE and RANDOM study follow-up completion, adherence, and weight loss among Non-Hispanic White and among those who identify to an ethnic and/or racial minoritized group. Quantitative analyses, however, do not make it possible to contextualize drivers that may influence relative preference, retention, and adherence. Using semi-structured interviews (Appendix A), we will explore the depth of personal beliefs and experiences, cultural contexts, social dynamics, social support systems, and household factors that may influence affect participants' preferences and sustained engagement. This knowledge will inform personalized behavior change strategies that are sensitive to the diverse needs of participants' social context.
Weight | Baseline, 6 Month, 12 Month
  Weight is measured using the Bluetooth enabled scales based on standard practices (e.g., empty pockets). Weight loss will be operationalized as the difference between weight at baseline, 6mo, and 12mo.

OTHER OUTCOMES:
Dietary intake and physical activity | Baseline, 6 Month, 12 Month
  We will leverage data conferred by the WW program to capture dietary intake and physical activity (type, duration and intensity) via the WW mobile app or online website.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Salvy, PhD, Principal Investigator — Cedars-Sinai Medical Center

IPD SHARING:
Plan to Share IPD: No